CLINICAL TRIAL: NCT07144839
Title: Clinical Utility of a Predictive Model of Placental Insufficiency
Brief Title: Placental Risk Assessment to CusTomize Individualized Pregnancy Care and Evaluation
Acronym: PRACTICE
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Karen Gibbins, Principal Investigator, Oregon Health and Science University
Other Study IDs: STUDY00026808; 1R01HD115604-01 (NIH)
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Stillbirth; Placental Insufficiency
MeSH Terms: conditions — Stillbirth; Placental Insufficiency | interventions — Parturition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma without DNA will be retained in the OHSU repository for potential future research.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort: Pregnant people age 15 and older, without known major fetal anatomic or genetic abnormalities, singleton gestation will be monitored via ultrasound and blood tests throughout pregnancy. Delivery data and neonatal outcomes will be collected. Data will be used to develop a predictive model of placental insufficiency.
  Interventions: Other: Data Collection Throughout Pregnancy and Delivery

INTERVENTIONS:
Other: Data Collection Throughout Pregnancy and Delivery — Participants will receive monitoring by ultrasound and blood tests at three time points during pregnancy, and delivery and neonatal data will be collected.

SUMMARY:
This is a prospective observational study with the goal of developing and assessing a predictive model of placental insufficiency.

DETAILED DESCRIPTION:
Pregnant study participants will be recruited and monitored throughout pregnancy with ultrasound and blood draws, and delivery and neonatal data up to 28 days following birth. This data will be used to develop a model to predict placental insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Age 15 or older
* No known major fetal anatomic or genetic abnormalities
* Singleton gestation
* Planning to deliver at Oregon Health & Science University
* Prior to 22 weeks' gestation

Exclusion Criteria:

* Decisional impairment
* Multiple gestation
* Known fetal growth restriction or major congenital anomaly
* Inability to consent
* Inability to attend study visits

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant people age 15 and older, parous and nulliparous, without known major fetal anatomic or genetic abnormalities. Participants must be pregnant with a singleton living gestation, less than 22 weeks' gestation at enrollment, and planning to deliver at Oregon Health & Science University.
Sampling Method: Non-Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with placental insufficiency composite | At time of delivery to 28 days following delivery
  The composite is made of the following: stillbirth and neonatal death, severe forms of hypertensive disease, placental abruption, birthweight below the 3rd percentile, umbilical cord arterial pH<7, and/or placental primary indication for delivery (FGR, oligohydramnios, abnormal fetal testing)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Gibbins, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States